CLINICAL TRIAL: NCT01906892
Title: Creative Practice as Mutual Recovery: Connecting Communities for Mental Health and Wellbeing
Brief Title: Creative Practice as Mutual Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Music (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AH/K003364/1
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Individuals Experiencing Mild or Moderate Mental Health Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1a (Experimental): 6 weeks of group drumming workshops
  Interventions: Other: Group drumming (participatory)
- 1b (Experimental): 6 weeks of group drumming workshops
  Interventions: Other: Group drumming (participatory)
- 2a (Experimental): 2 weeks of active group drumming followed by 2 weeks of control activity involving a literary-based activity
  Interventions: Other: Group drumming (participatory); Other: Comparative activity
- 2b (Active Comparator): 2 weeks of the literary-based comparative activity followed by 2 weeks of watching live group drumming
  Interventions: Other: Group drumming (live); Other: Comparative activity
- 2c (Active Comparator): 2 weeks of listening to live group drumming followed by 2 weeks of listening to recordings of group drumming
  Interventions: Other: Group drumming (live); Other: Group drumming (recorded)
- 2d (Active Comparator): 2 weeks of listening to recorded group drumming followed by 2 weeks of participation in group drumming
  Interventions: Other: Group drumming (participatory); Other: Group drumming (recorded)
- 3a (Experimental): 10 weeks of participatory group drumming workshops
  Interventions: Other: Group drumming (participatory)
- 3b (Active Comparator): 10 weeks of engagement with other non-musical social activities
  Interventions: Other: Group drumming (participatory)

INTERVENTIONS:
Other: Group drumming (participatory) — Active participation in group drumming workshops
  Arms: 1a; 1b; 2a; 2d; 3a; 3b
Other: Group drumming (live) — Listening to live performances of group drumming
  Arms: 2b; 2c
Other: Group drumming (recorded) — Listening to recorded performances of group drumming
  Arms: 2c; 2d
Other: Comparative activity — Taking part in a literary-based activity
  Arms: 2a; 2b

SUMMARY:
This study explores the hypothesis that mental health service users, their carers and musicians can - through the creative act of music learning and performing - mutually enhance wellbeing through the development of more meaningful and resilient lives. The project seeks to explore three interconnected issues: (i) the extent to which music learning and performing provides a forum for 'mutual recovery' among adult mental health service users, their formal/informal carers, and musicians, (ii) the characteristic features of 'mutual recovery' through music, and (iii) the underlying mechanisms of such 'mutual recovery'.

The study will consist of three different stages. Stages 1 and 2 will examine the effect of a variety of group activities - including participatory music, listening to live music, listening to recorded music and a non-music control - on psychological scales, saliva samples of stress hormones and cytokines, and subjective experience to see which provide the most relaxing, sociable and supportive environments for mutual recovery. Stage 3 will explore the impact of musical interventions over longer periods of time.

A systematic review we have just carried out has revealed a major gap in research comparing different music interventions and testing the effects of different lengths of interventions. As a result, our study should help us answer the following questions:

* Which aspect(s) of music can contribute to mutual recovery?
* Do carers, patients and musicians all respond to the same activities, or do some musical activities suit certain groups more than others?
* Do carers, patients and musicians all recover at the same rate?
* What length of intervention is most effective?

If certain interventions are found to produce stronger results than others, these results could help guide community groups and healthcare settings in their design of music activities and have implications for the spending of arts-in-health budgets.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of either gender and over the age of 18 who are experiencing mild or moderate mental health issues including but not limited to: stress, anxiety, depression etc.
* Individuals of either gender and over the age of 18 who formally or informally care for mental health service users.
* Musicians who are professional workshop leaders and music students training to be professional musicians.

Exclusion Criteria:

* Serious mental health problems which might

  1. prevent an individual from giving informed consent
  2. cause the individual to be a disruption to other participants
* Individuals for whom the music activity might conflict with other routine care.
* Individuals with gum disease which would invalidate saliva samples.
* Total deafness or severely impaired hearing.
* Musicians or music students who apply to participate in the project but who are not deemed to have sufficient experience or expertise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Well-being Scale | Change from baseline (recorded in the week prior to participation in either 6 or 10 weeks of music interventions) to the end of participation in the music interventions

SECONDARY OUTCOMES:
Secker's 'Measure of social inclusion for arts and mental health project participants' | Change from baseline (recorded in the week prior to participation in either 6 or 10 weeks of music interventions) to (a) the end of participation in the music interventions, and (b) 3 months after the end of music interventions
Connor-Davidson Resilience Scale (CD-RISC) | Change from baseline (recorded in the week prior to participation in either 6 or 10 weeks of music interventions) to (a) the end of participation in the music interventions, and (b) 3 months after the end of music interventions
Hospital Anxiety and Depression Scale | Change from baseline (recorded in the week prior to participation in either 6 or 10 weeks of music interventions) to (a) the end of participation in the music interventions, and (b) 3 months after the end of music interventions
Saliva levels of cortisol | Change from baseline (taken immediately before the music intervention) when measured immediately following the 60 or 90 minute music intervention session
Blood pressure | Change from baseline (taken immediately before the music intervention) when measured immediately following the 60 or 90 minute music intervention session
Saliva levels of salivary immunoglobulin A | Change from baseline (taken immediately before the music intervention) when measured immediately following the 60 or 90 minute music intervention session
Saliva levels of interleukins including IL6 | Change from baseline (taken immediately before the music intervention) when measured immediately following the 60 or 90 minute music intervention session
Heart rate | Change from baseline (taken immediately before the music intervention) when measured immediately following the 60 or 90 minute music intervention session

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Williamon, PhD, Principal Investigator — Royal College of Music
Locations (1):
- Centre for Performance Science, Royal College of Music, London, United Kingdom

REFERENCES:
- [Derived] Fancourt D, Perkins R, Ascenso S, Carvalho LA, Steptoe A, Williamon A. Effects of Group Drumming Interventions on Anxiety, Depression, Social Resilience and Inflammatory Immune Response among Mental Health Service Users. PLoS One. 2016 Mar 14;11(3):e0151136. doi: 10.1371/journal.pone.0151136. eCollection 2016. PMID 26974430
- [Derived] Fancourt D, Perkins R, Ascenso S, Atkins L, Kilfeather S, Carvalho L, Steptoe A, Williamon A. Group Drumming Modulates Cytokine Response in Mental Health Services Users: A Preliminary Study. Psychother Psychosom. 2016;85(1):53-5. doi: 10.1159/000431257. Epub 2015 Nov 27. No abstract available. PMID 26610172